CLINICAL TRIAL: NCT01726192
Title: Comparison of Ultrasound Hydrolocalization Technique Versus Neurostimulation for Placement of Continuous Femoral Catheters.
Brief Title: Comparison of Two Techniques for Placement of Perineural Femoral Catheters.
Acronym: HLOCSTIM2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Sidiropoulou Tatiana, Lecturer in Anesthesiology, University of Athens, Attikon Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HLOCSTIM2
Record Dates: First submitted 2012-11-09; First posted 2012-11-14 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Postoperative Pain; Anterior Cruciate Ligament Reconstruction
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HLOC (Active Comparator): Placement of a femoral catheter with the hydrolocalization technique
  Interventions: Procedure: Placement of a femoral catheter with the hydrolocalization technique
- NS (Active Comparator): Placement of a femoral neurostimulating catheter
  Interventions: Procedure: Placement of a femoral neurostimulating catheter

INTERVENTIONS:
Procedure: Placement of a femoral catheter with the hydrolocalization technique — Placement of femoral nerve catheter with the hydrolocalization technique, using ropivacaine 0.6%
  Other Names: Placement of femoral nerve catheter with the hydrolocalization technique, using ropivacaine 0.6%
  Arms: HLOC
Procedure: Placement of a femoral neurostimulating catheter
  Arms: NS

SUMMARY:
The purpose of this study is to assess the efficacy of the hydrolocalization technique for placement of femoral perineural catheters in comparison with stimulating catheters. A non inferiority trial.

DETAILED DESCRIPTION:
The investigators will randomize patients that will undergo anterior cruciate ligament reconstruction.

Each patient will receive a subgluteal single shot nerve block and a continuous femoral nerve block with placement of a catheter either with the hydrolocalization technique (group HLOC) or a neurostimulating catheter (group NS).

ELIGIBILITY:
Inclusion Criteria:

* adults
* BMI less than 30

Exclusion Criteria:

* known allergies to local anesthetics or other drugs used
* patient refusal
* any local or systemic contraindication to the use of popliteal block

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
local anesthetic consumption | 36 hours postoperatively

SECONDARY OUTCOMES:
Pain scores with a VAS scale | 36 hours postoperatively

OTHER OUTCOMES:
incidence of side effects, consumption of iv analgesics | 36 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana F Sidiropoulou, MD, PhD, Principal Investigator — Attikon Hospital; Theodosios Saranteas, MD, PhD, Principal Investigator — Attikon Hospital; Mario Dauri, MD, Principal Investigator — Policlinico Tor Vergata
Locations (2):
- Attikon Hospital, Athens, Greece
- Policlinico Tor Vergata, Rome, Italy

REFERENCES:
- [Background] Saranteas T, Adoni A, Sidiropoulou T, Paraskeuopoulos T, Kostopanagiotou G. Combined ultrasound imaging and hydrolocalization technique for accurate placement of perineural catheters. Br J Anaesth. 2011 Dec;107(6):1008-9. doi: 10.1093/bja/aer375. No abstract available. PMID 22088876